CLINICAL TRIAL: NCT00754091
Title: Retention of an Orally Administered Investigational Device in the Oropharynx of Healthy Human Male Volunteers
Brief Title: Evaluate Retention of an Orally Administered Device Using Gamma Scintigraphy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008046
Record Dates: First submitted 2008-07-09; First posted 2008-09-17 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Polymer based lubricating liquid

INTERVENTIONS:
Device: Polymer based lubricating liquid — three sprays of radiolabeled polymer blend of carboxymethylcellulose, polyoxyl 40 stearate, and polyethylene oxide that coats and protects the mucus membrane

SUMMARY:
Single usage, open label study in 16 adult healthy males. Eligible subjects will receive a single usage of the investigational device. Retention of the radiolabeled device will be monitored using gamma scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Refrain from nasal, throat, or lung inhalants and exercise for 24 hour prior to the test
* Are able to tolerate the procedure and
* Be generally healthy

Exclusion Criteria:

* Have history of allergy or hypersensitivity to the study ingredients
* Major diseases
* Taking medication regularly
* Radiation exposure recently

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve for the percent of the mucoadhesive liquid retained in the oropharynx | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Doll, PhD, RPh, Principal Investigator — Scintipharma, Inc
Locations (1):
- Walter J Doll, PhD, RPh, Lexington, Kentucky, United States